CLINICAL TRIAL: NCT06091423
Title: XELOX Combined With Fruquintinib and Sintilimab Regimen Conversion Therapy for Gastric Cancer/Gastroesophageal Junction Adenocarcinoma Only With Liver and/or Retroperitoneal Lymph Node Metastasis, a Prospective Single-arm, Multicenter Study ( FISSION Study )
Brief Title: XELOX Combined With Fruquintinib and Sintilimab Regimen Conversion Therapy for Gastric Cancer/Gastroesophageal Junction Adenocarcinoma Only With Liver and/or Retroperitoneal Lymph Node Metastasis, a Prospective Single-arm, Multicenter Study
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Xiaofeng Chen (Other)
Responsible Party: Sponsor-Investigator, Xiaofeng Chen, professor, The First Affiliated Hospital with Nanjing Medical University
Organization: The First Affiliated Hospital with Nanjing Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Fission
Record Dates: First submitted 2023-10-10; First posted 2023-10-19 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Gastric Cancer/Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Stomach Neoplasms | interventions — HMPL-013; sintilimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): XELOX combined with Fruquintinib and Sintilimab
  Interventions: Drug: XELOX combined with Fruquintinib and Sintilimab

INTERVENTIONS:
Drug: XELOX combined with Fruquintinib and Sintilimab — XELOX:Capecitabine：800mg/m2, po, bid, d1-14。Oxaliplatin：130mg/m2，ivgtt 2-6h，d1，q3w; Fruquintinib: 5 mg/d，qd po，d1-14，q3w; Sintilimab: 200mg d1, q3w

SUMMARY:
Gastric cancer is the third leading cause of morbidity and mortality among malignant tumors in China, and less than 30% of patients can be cured by surgery. Liver metastasis, retroperitoneal lymph node metastasis and peritoneal metastasis are the most common metastatic sites of gastric cancer, which are also the important causes of death. Improve the conversion of oligonucleotides transfer patients resection rate, prolonged progression-free survival of these patients, is an important direction to improve survival of patients with advanced gastric cancer;

This study was a prospective, single-arm, multi-center clinical study. We plan to treat patients with gastric cancer/gastroesophageal junction adenocarcinoma with liver and/or retroperitoneal lymph node metastasis only with XELOX regimen + fruquinitinib + sintilimab for 4-6 cycles before surgery/ablation conversion therapy to achieve tumor-free status as far as possible. To explore the value of conversion therapy in patients with intrahepatic oligometastasis of gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18-75 years of age;
2. Understand the steps and content, and written informed consent signed voluntarily;
3. Is confirmed by histopathology and/or cytology her2-negative or HER2 status unknown late recurrence or stomach esophagus stomach/integration of adenocarcinoma;
4. In this research to define transfer of oligonucleotides definition: the primary lesion and regional lymph node metastasis of process to determine the surgeon can be cut or boundary can be cut, only intrahepatic metastasis and distant metastasis (metastases number 5 or less, a single lesion or less 5 cm in diameter.) And or retroperitoneal lymph node metastasis (16a2,16b1,16a1,16b2 metastasis), no other distant metastasis;
5. At least one measurable lesion according to RECIST 1.1 criteria;
6. No previous treatment with VEGFR-targeted drugs and PD-1/PD-L1 monoclonal antibodies. Patients who had relapsed more than 6 months after the completion of postoperative adjuvant chemotherapy with platinum or paclitaxel or fluorouracil and had no grade 2 or higher toxicity were eligible for enrollment.
7. ECOG PS score: 0-1;
8. Expected survival time ≥3 months;
9. The main viscera function is good, namely into groups of related within 14 days before check index meet the following requirements:

(1) hemoglobin ≥80 g/L; (2) neutrophil count >1.5×109/L; (3) platelet count ≥80×109/L; (4) Total bilirubin ≤2.5×ULN (upper limit of normal); (5) serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) ≤5×ULN; (6) the endogenous creatinine clearance or 60 ml/min (Cockcroft - Gault formula); (7) Echocardiography: left ventricular ejection fraction (LVEF)≥50%; (8) Thyroid function indexes: thyroid stimulating hormone (TSH) and free thyroxine (FT3/FT4) were in the normal range or only mildly abnormal, without related clinical symptoms; (9) A body weight of 40 kg or more, or a BMI > 18.5;

Exclusion Criteria:

1. Patients with other malignant tumors in the past or at the same time, but have been cured of early tumors, including basal cell carcinoma of the skin and carcinoma in situ of the cervix, stage I lung cancer, stage I colorectal cancer and other tumors that do not affect the patient's life in the short term according to the investigator's judgment can be excluded;
2. Participated in other drug clinical trials within four weeks;
3. Multiple factors affecting oral medication (such as inability to swallow, chronic diarrhea and intestinal obstruction);
4. Patients with a history of bleeding and any bleeding events of CTCAE5.0 grade 3 or higher within 4 weeks before screening;
5. Metastasis in other distant sites, including but not limited to lung metastasis, brain metastasis, bone metastasis, distant lymph node metastasis, and peritoneal metastasis;
6. Patients with hypertension not well controlled by single antihypertensive medication (systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg); Patients with a history of unstable angina; Newly diagnosed angina pectoris within 3 months before screening or myocardial infarction within 6 months before screening; Arrhythmias (including QTcF ≥450 ms in men and ≥470 ms in women) required long-term use of antiarrhythmic drugs and New York Heart Association (NYHA) grade ≥II cardiac dysfunction;
7. Long-term unhealed wounds or incompletely healed fractures;
8. Imaging shows that the tumor has invaded the important blood vessels or the investigator judges that the patient's tumor has a high possibility of invading the important blood vessels during the treatment and causing fatal hemorrhage;
9. Abnormal coagulation function, with bleeding tendency (14 days before enrollment must meet: INR in the normal range without anticoagulant or clinically insignificant abnormality); Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin, or their analogues; International standardization in prothrombin time ratio (INR) under the premise of 1.5 or less, allowing purpose to prevent the use of low-dose warfarin (1 mg orally, once per day) or low-dose aspirin (amount does not exceed 100 mg daily);
10. Occurrence of arterial/venous thrombosis events within 6 months before screening, such as cerebrovascular accident (including transient ischemic attack), deep vein thrombosis (except for venous thrombosis caused by venous catheterization due to previous chemotherapy and judged by investigators to be cured), and pulmonary embolism;
11. Urine routine showed urine protein ≥++ and confirmed 24-hour urine protein quantitation >1.0 g;
12. Previous use of immune-targeted therapy drugs;
13. Have a history of immunodeficiency or other acquired or congenital immunodeficiency diseases, or have a history of organ transplantation;
14. Patients with infectious pneumonia, non-infectious pneumonia, interstitial pneumonia and other patients requiring corticosteroids;
15. A history of severe chronic autoimmune diseases, such as systemic lupus erythematosus; He had a history of inflammatory bowel disease such as ulcerative enteritis, Crohn's disease, and a history of chronic diarrhea such as irritable bowel syndrome. A history of sarcoidosis or tuberculosis; Patients with a history of active hepatitis B or C, and HIV infection; Good control of severe autoimmune disease, such as dermatitis, arthritis, psoriasis, etc can be into the group. Patients with hepatitis B virus titer <1000copy/ml were eligible for enrollment.
16. Patients with hypersensitivity to human or murine monoclonal antibodies;
17. Have a history of psychotropic drug abuse and cannot quit or have mental disorders;
18. Patients who do not follow the doctor's advice, do not follow the prescribed medication, or have incomplete data, which may affect the efficacy or safety judgment;
19. Concomitant diseases that, in the judgment of the investigator, seriously compromise patient safety or interfere with patient completion of the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2025-11-25 (Estimated); Study Completion 2026-11-25 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year]
  Time from randomization to disease progression or death from any cause

SECONDARY OUTCOMES:
Overall survival (OS） | from randomization until death due to any cause, assessed up to 3 year
  Overall survival means any reason from patients into groups to the date of death
Objective response rate (ORR) | Time Frame: from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  the proportion of patients with complete response or partial response, using RECIST v 1.1.
Disease Control Rate (DCR) | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  the proportion of patients with complete response, partial response or stable disease, using RECIST v 1.1.
Duration of Response (DOR) | from randomization up to progressive disease or EOT due to any cause, assessed up to 2 year
  Cancer for the first time that assessment for CR or PR to the first evaluation for PD or any cause the time of death.
translational rate | 2-3 months
  It refers to the proportion of all enrolled patients who underwent radical surgery/ablation therapy after medical treatment.
Adverse event (AEs) | 2 years
  Toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0. The number of Participants with adverse events will be recorded at each treatment visit.

CONTACTS AND LOCATIONS:
Locations (1):
- Jiangsu Province Hospita, Nanjin, China

IPD SHARING:
Plan to Share IPD: Undecided